CLINICAL TRIAL: NCT05754268
Title: Establishment, Verification and Clinical Application of Chinese Version of Surgical Risk Assessment System
Acronym: CSRAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: luyun (Other)
Responsible Party: Sponsor-Investigator, luyun, Chief physician, The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Other Study IDs: CSRAS
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Risk Assessment; Risk Factors; Machine Learning; Artificial Intelligence; Postoperative Complications; Operative Surgical Procedure
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese version of Surgical risk Assessment system Group: This group of patients used the Chinese version of the surgical risk assessment system to evaluate the complications.
  Interventions: Procedure: Chinese version of the surgical risk assessment system

INTERVENTIONS:
Procedure: Chinese version of the surgical risk assessment system — There is no need to interfere with the patient. Investigators can observe the outcome after using the system for evaluation.

SUMMARY:
The goal of this observational study is to establish and verify the Chinese version of surgical risk assessment system and explore its clinical application. The main questions it aims to answer are: The process of establishing a Chinese version of surgical risk assessment system; What is the accuracy of the system; How can the system be used in clinic; How does this system compare with other systems (such as NSQIP). Participants will comprehensively collect the general information, examination and pathological information of the patients, using machine learning and artificial intelligence methods for data processing. Finally, the Chinese version of the surgical risk assessment system will be established. After the system is established, investigators will evaluate the accuracy of the system and compare it with other related systems.

DETAILED DESCRIPTION:
The research process is as follows:

1. Determine the collection index and the complications to be evaluated, and retrospectively collect the preoperative clinical data (including preoperative medical records, examination and examination results) of patients with postoperative complications of gastric and colorectal cancer in our hospital in the past ten years. Preliminary construction of surgical risk assessment system (gastrointestinal surgery)
2. Retrospective or prospective collection of gastric cancer and colorectal surgery cases (not included in the system)
3. The occurrence of postoperative complications was observed until 1 month after discharge. Compare the evaluation results of the system with the actual situation and feedback to further improve the system.
4. The same batch of patient data can be input into NSQIP to re-evaluate and predict the occurrence of patient complications, and then compare the results of the two systems.
5. The incidence of postoperative complications (number of cases and accuracy) of the two groups were counted respectively, and the accuracy and practicability of the evaluation of the two systems were compared to further improve the system.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative colonoscopy and biopsy confirmed gastric and colorectal cancer.
* Laparotomy or laparoscopic radical resection of gastric or colorectal cancer.
* No postoperative complications such as pneumonia, venous thrombosis, cardiovascular and cerebrovascular accidents occurred before operation.
* There was no serious organ dysfunction before operation.
* Complete auxiliary examination and the availability of examination and examination data were carried out before operation.

Exclusion Criteria:

* Complicated with malignant tumors of other organs.
* Unresectable tumors.
* Distant metastasis.
* Severe organ system dysfunction before operation.
* Patients with non-operative treatment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mainly collect the patients who were diagnosed as gastric cancer or colorectal cancer and received a single limited period of surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of complications | Within one month after the operation
  The following complications occurred or did not occur in the patient: death, cardio-cerebrovascular accident, pneumonia, lower extremity deep venous thrombosis, anastomotic fistula, incision infection, intrabody periorgan infection, systemic septicemia, urinary system infection, renal insufficiency / failure, unplanned reoperation, intestinal obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Yun, Doctor, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Yiheng Ju, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided